CLINICAL TRIAL: NCT02052687
Title: A First-in-human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LFX453, After Multiple Topical Applications in Healthy Volunteers.
Brief Title: A First-in-human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LFX453
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: CLFX453X2101; 2013-002344-84 (EudraCT Number)
Record Dates: First submitted 2014-01-15; First posted 2014-02-03 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Healthy volunteer
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1: LFX453/placebo (Experimental): once daily: LFX453 cream 1 high dose / LFX453 cream 1 low dose /Placebo 1 / LFX453 cream 2 high dose / LFX453 cream 2 low dose / Placebo 2
  Interventions: Drug: LFX453 H1; Drug: LFX453 L1; Drug: LFX453 H2; Drug: LFX453 L2; Drug: Placebo 1; Drug: Placebo 2
- Part 2 groupA: LFX453/placebo (Experimental): once daily: LFX453 cream 1 / Placebo 1
  Interventions: Drug: LFX453 H1; Drug: LFX453 L1; Drug: LFX453 H2; Drug: LFX453 L2; Drug: Placebo 1; Drug: Placebo 2
- Part 2 groupB: LFX453/placebo (Experimental): once daily: LFX453 cream 2 / Placebo 2
  Interventions: Drug: LFX453 H1; Drug: LFX453 L1; Drug: LFX453 H2; Drug: LFX453 L2; Drug: Placebo 1; Drug: Placebo 2
- Part 2 groupC: LFX453/LFX453 (Experimental): once daily: LFX453 cream 1 / LFX453 cream 2
  Interventions: Drug: LFX453 H1; Drug: LFX453 L1; Drug: LFX453 H2; Drug: LFX453 L2
- Part 2 groupD: Imiquimod (Other): once daily: imiquimod cream
  Interventions: Drug: Imiquimod
- Part 3: LFX453/placebo (Experimental): twice daily: LFX453 cream 1 high dose / LFX453 cream 1 low dose /Placebo 1 / LFX453 cream 2 high dose / LFX453 cream 2 low dose / Placebo 2
  Interventions: Drug: LFX453 H1; Drug: LFX453 L1; Drug: LFX453 H2; Drug: LFX453 L2; Drug: Placebo 1; Drug: Placebo 2

INTERVENTIONS:
Drug: LFX453 H1 — LFX453 high dose cream 1
  Arms: Part 1: LFX453/placebo; Part 2 groupA: LFX453/placebo; Part 2 groupB: LFX453/placebo; Part 2 groupC: LFX453/LFX453; Part 3: LFX453/placebo
Drug: LFX453 L1 — LFX453 low dose cream 1
  Arms: Part 1: LFX453/placebo; Part 2 groupA: LFX453/placebo; Part 2 groupB: LFX453/placebo; Part 2 groupC: LFX453/LFX453; Part 3: LFX453/placebo
Drug: LFX453 H2 — LFX453 high dose cream 2
  Arms: Part 1: LFX453/placebo; Part 2 groupA: LFX453/placebo; Part 2 groupB: LFX453/placebo; Part 2 groupC: LFX453/LFX453; Part 3: LFX453/placebo
Drug: LFX453 L2 — LFX453 low dose cream 2
  Arms: Part 1: LFX453/placebo; Part 2 groupA: LFX453/placebo; Part 2 groupB: LFX453/placebo; Part 2 groupC: LFX453/LFX453; Part 3: LFX453/placebo
Drug: Imiquimod — Imiquimod cream
  Arms: Part 2 groupD: Imiquimod
Drug: Placebo 1 — Placebo cream 1
  Arms: Part 1: LFX453/placebo; Part 2 groupA: LFX453/placebo; Part 2 groupB: LFX453/placebo; Part 3: LFX453/placebo
Drug: Placebo 2 — Placebo cream 2
  Arms: Part 1: LFX453/placebo; Part 2 groupA: LFX453/placebo; Part 2 groupB: LFX453/placebo; Part 3: LFX453/placebo

SUMMARY:
The purpose of this first-in human study is to demonstrate systemic and local tolerability and investigate pharmacokinetics of LFX453 after multiple topical applications in healthy subjects.

The current study has been designed with three distinct parts. Part 1 focuses on safety and tolerability of once daily application on the back, prior to moving forward and assessing the safety and tolerability in more sensitive treatment areas in Part 2 or twice daily application in Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects of non-childbearing potential, 18 to 65 years of age inclusive (at the time of the screening visit), and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Male subjects must agree to total abstinence from male:female intercourse or agree to use a condom during drug dosing and for four weeks after dosing has stopped.

Exclusion Criteria:

* History of serious allergic reaction to any drug.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* History of any atopic dermatitis (only within the last 2 years), autoimmune disease, psoriasis or erythema multiforme.
* Presence of skin disease (e.g. warts) or skin features on treatment areas that may affect local tolerability or the ability of the investigator to evaluate local tolerability.
* History of heart failure, left ventricular dysfunction or known family history or known presence of long QT syndrome.
* A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening or baseline:

  * 2nd or 3rd degree AV-block
  * PR > 200 msec
  * QRS complex > 120 msec
  * QTcF > 450 msec (males)
  * QTcF > 460 msec (females)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
General safety (number of subjects with adverse events) | 14 days
  Summarized statistics on adverse events will be reported under categories such as total adverse events, serious adverse events and death.
Local skin tolerability (tolerability score) | 14 days
  Summarized statistics on 5-point scale tolerability scores over 14 days of treatment.

SECONDARY OUTCOMES:
All parts: Amount (ng/mL) of LFX453 in plasma | 14 days
  Evaluate systemic steady state pharmacokinetics in human after topical administration of LFX453.
Part 1 and 2: LFX453 concentrations (ng/g) in the skin | Day 14 and between days 18-21
  LFX453 analyzed in skin.
All parts: LFX453 concentration (ng/mL) in urine | Day 14
  LFX453 analyzed in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Mid Glamorgan, United Kingdom